CLINICAL TRIAL: NCT04511325
Title: Effects of White Potato Consumption on Measures of Cardiometabolic Health in Individuals With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Neda Akhavan, Dr. Neda S. Akhavan, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 00000498
Record Dates: First submitted 2020-07-30; First posted 2020-08-13 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Type2 Diabetes; Cardiometabolic Syndrome; Arterial Stiffness; Overweight and Obesity
Keywords: Functional Foods; Chronic Diseases; Carbohydrates; Endothelial Dysfunction; Cardiometabolic Health
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Chronic Disease

STUDY DESIGN:
Intervention Model Description: For this randomized cross-over study, participants (45-80 y, BMI 25-35 kg/m2, fasting blood glucose >126 g/dL, HbA1c 6.5-9%, non-frequent white potato consumption of <2 servings per week) will be randomly assigned to receive pre-prepared baked white potato (100g cooked with skin; 100kcals) or a calorie-matched refined grain (75g cooked long-grain white rice; control) daily for each or two 12-week treatment periods, separated by a 2-week washout. Randomization of participants in the potato or the calorie-matched refined grain group will be done during the screening visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato Regimen Arm (Other): All participants will be randomly assigned to receive the potato regimen daily for the 12-week treatment period, separated by a 2-week washout.The potato regimen (75 grams of baked white russet potato with the skin) and refined grain (100 grams of long grain white rice) regimen will be matched for calories, carbohydrate and fat content and will both contribute to approximately 100 kilocalories, 22g carbohydrates, and 0.2g of fat. In order to increase participants' compliance, they will be informed of a variety of ways to consume their regimen. The rationale for choosing this amount of potato and rice regimen is based on the common practice of carbohydrate counting practiced by dietitians and diabetes educators in clinical settings, where 45-60 g of carbohydrates should be consumed at each meal and 15-20 g of carbohydrates can be consumed at each snack throughout the day.
  Interventions: Other: Potato Regimen
- Refined Grain Regimen Arm (Other): All participants will be randomly assigned to the calorie-matched refined grain daily for the 12-week treatment period, separated by a 2-week washout.The refined grain (100 grams of long grain white rice) regimen will be matched to the potato regimen for calories, carbohydrate and fat content and will both contribute to approximately 100 kilocalories, 22g carbohydrates, and 0.2g of fat. In order to increase participants' compliance, they will be informed of a variety of ways to consume their regimen. The rationale for choosing this amount of potato and rice regimen is based on the common practice of carbohydrate counting practiced by dietitians and diabetes educators in clinical settings, where 45-60 g of carbohydrates should be consumed at each meal and 15-20 g of carbohydrates can be consumed at each snack throughout the day. Long-grain boiled white rice also has a similar glycemic index to that of a baked white potato.
  Interventions: Other: Refined Grain Regimen

INTERVENTIONS:
Other: Potato Regimen — 100 grams cooked white russet potato with the skin
  Arms: Potato Regimen Arm
Other: Refined Grain Regimen — 75 grams of cooked long-grain white rice
  Arms: Refined Grain Regimen Arm

SUMMARY:
The investigators are examining the effects of potato consumption on indices of glycemic control and cardiovascular health in overweight and obese individuals with type two diabetes mellitus (T2D) to provide feasible and effective dietary ways for individuals to enhance their quality of life. The overall objective of this crossover study is to collect data regarding the effects of potato consumption on indices of glycemic control and cardiovascular health among overweight and obese individuals with T2D. The central hypothesis of this crossover study is that the daily consumption of 100 g white potato for 12 weeks will contribute to improvements in glycemic control, reductions in inflammation, and improvements in blood lipids and vascular function in overweight and obese individuals with T2D compared to a macronutrient-matched refined grain (75 g cooked long-grain white rice) for 12 weeks (with a 2 week washout period between interventions).

Specific Aim) The assessment of blood glucose control, vascular function, body composition and overall cardiovascular risk after consumption of potatoes (100g/d for 12 weeks) in individuals with T2D compared to a calorie matched refined grain at the initial baseline visit as well as the 6-, and 12-week study visits (for each 12-week intervention period).

This aim will assess changed in blood glucose, insulin, HbA1c, HOMA-IR, and HOMA-β as well as the following:

1. blood pressure (BP)
2. markers of endothelial function [flow-mediated dilation (FMD), pulse wave velocity (PWV), and endothelin-1 (ET-1)]
3. markers of inflammation (C-reactive protein)
4. body composition via bioelectrical impedance (BIA), lean mass and fat mass assessment
5. lipid profiles, consisting of total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and oxidized LDL (Ox-LDL). Atherogenic risk ratios (TC/HDL-C, LDL-C/HDL-C, HDL-C/LDL-C) will also be assessed
6. anthropometrics [weight, height, waist circumference (WC), hip circumference (HC), waist-to-hip ratio (WC/HC)]

DETAILED DESCRIPTION:
A total of 50 men and postmenopausal women between the ages of 45 and 80 who have T2D will be recruited for this study. Participants with T2D will be recruited from Tallahassee, FL and surrounding areas through campus and community advertisements through flyers, newspaper articles, and public events. After an initial telephone screening, all participants will be requested to report to the clinical area of the Sandels building at FSU (study site) for their first on-site visit (and all visits if the participant qualifies). On the first visit (screening), the potential participants will be provided with verbal and written explanation of the project and will have any questions regarding the study answered by trained research personnel during the informed consent process. Then the individual will be asked to sign an informed consent form, followed by a medical history questionnaire to confirm their diabetic state, and measurements of their fasting blood glucose levels and HbA1c will also be done to assess any changes that may occur throughout the study. Anthropometrics will be measured and questions on medical history and medication use will be asked during the screening visit to confirm eligibility. Randomization of participants in the potato or the calorie-matched refined grain group will be done after the screening visit and following completion of a Seven-Day Food Frequency Questionnaire (FFQ), which will indicate if individuals frequently consume potatoes. If participants are considered "non-frequent" white potato consumers (<2 servings per week), they will be included in this study and asked to come for following visits, additionally during this visit participants will be familiarized with vascular assessments prior to their baseline appointment. On the second (baseline) visit participants will be randomly assigned to one of two groups: 1) 100 g cooked white potato or 2) 75 g calorie-matched cooked refined grain (cooked long-grain white rice) daily for 12 weeks following a 2-week washout period prior to the other intervention group (a total of 26 weeks upon completion of the study). Study foods will be prepared at the Florida State University Metabolic Kitchen and Diet Assessment Lab following SafeStaff Foodhandler Training, an approved Florida foodhandler program, protocols for preparation, storage and handling. At the baseline visit participants will be asked to come fasted; BP and vascular function will be measured followed by blood draw, anthropometrics, body composition (via BIA), and a physical activity questionnaire will be administered. Participants will be provided with their assigned dietary regimen and will receive instructions on how to fill out daily diaries for their dietary regimen and will be given three-day food records to bring back for their subsequent visits to assess typical intake throughout the study. BP, vascular function, blood draw, and anthropometric, body composition, diet, and physical activity assessments will be repeated at 6-, and 12-week visits for both intervention periods with a 2-week washout between each intervention period (for a total of 5 study visits). After the 2-week washout period, participants will be asked to come to the study site, to receive the other intervention group and be given instruction on their new dietary regimen. Participants will be asked to come to the study site on a bi-weekly basis to pick up potato and white rice regimen, which can be stored in the freezer/refrigerator prior to consumption. Additionally, participants will be given portioned cooked rice to take home with them for the long-grain white rice regimen. All cardiovascular measurements will be performed between 7:00-10:00 A.M., in a quiet temperature-controlled room after an overnight fast and 12 hours after the abstinence of caffeine and/or 24 hours after the last bout of moderate to heavy physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* Overweight or obese individuals (BMI of 25-40 kg/m2),
* Individuals diagnosed type 2 diabetes.
* Individuals considered non-frequent potato consumers (< 2 serving of potatoes a week).

Exclusion Criteria:

* Individuals taking insulin
* Individuals diagnosed with CVD
* Individuals with uncontrolled hypertension (≥ 160/100 mmHg)
* Individuals with other active chronic diseases (cancer, asthma, glaucoma, thyroid, kidney, liver and pancreatic disease)
* Women who are pregnant/pre/perimenopausal, or on hormone replacement therapy
* Individuals with fasting blood glucose levels ≥ 200 mg/dL and HbA1c ≥ 9.0 %.
* Individuals participating in a weight loss program
* Individuals who are heavy smokers (> 20 cigarettes per day)
* Individuals who are heavy drinkers (> 12 alcoholic drinks per week)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-27 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on glucose in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in blood glucose from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on insulin in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in insulin from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on insulin resistance and insulin sensitivity in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in HOMA-IR and HOMA-β from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on hemoglobin A1c (HbA1c) in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in HbA1c from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on lipid profile in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in total cholesterol (TC), triglycerides (TG), high density lipoprotein-cholesterol (HDL-C), low density lipoprotein-cholesterol (LDL-C), oxidized-LDL (Ox-LDL) as well as atherogenic risk ratios (TC/HDL-C, LDL-C/HDL-C, HDL-C/LDL-C), from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on flow-mediated dilation (FMD) in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in flow-mediated dilation (FMD) from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period)on markers on inflammation/adhesion molecules in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in C-reactive protein and endothelin-1 (ET-1) from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on pulse wave velocity (PWV) in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in pulse wave velocity (PWV) from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.

SECONDARY OUTCOMES:
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on body composition in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes body composition via biolelectrical impedance (BIA), including lean mass and fat mass from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on BMI in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in BMI (weight and height) from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.
The effects of daily white potato versus white rice consumption for 12 weeks (each intervention for 12 weeks with a 2-week washout period) on waist-to-hip ratio in individuals with type 2 diabetes mellitus. | 26 weeks
  To examine changes in waist-to-hip ratio (waist and hip circumference) from Baseline, 6-week, and 12-week study visits (for each treatment period) in a total of 50 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Neda S Akhavan, PhD, Principal Investigator — Florida State University
Locations (1):
- Sandels Building, Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data collected in hard copy will be securely stored in a filing cabinet in our laboratory (Sandels 314). The data will only be accessible to the PI by key. De-identified data that is collected in soft copy will be stored on the PI's password protected computer. The data will be linked to subjects via encrypted codes to ensure their protection and confidentiality; the codes will not include HIPPA identifiers, such as initials, date of birth, etc. The encryption code for participants will be kept on the PI's computer; no other staff will have access to the encryption code. All data transferred from computer to computer will only be in the encrypted form. If identifiers are removed from the identifiable private information that are collected during this research, that information or those samples could be used for future research studies or distributed to other investigators for future research studies without additional informed consent.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data collection will be available once the participant has come in for their study visit and will be available for up to 10 years since the study has began unless otherwise extended.
Access Criteria: Only CITI trained and FSU trained research personnel will have access to data for the study following all University IRB guidelines. Research staff will be trained on the importance of participant confidentiality. Efforts will be made to limit the use and disclosure of personal information, including research study and medical records, to people who need to review this information. Data will be stored on the PI's password protected computer. Data will be stored until all analyses and reports are completed. Upon completion, data will be moved to the PI's password-protected computer for long-term storage. The PI will be responsible for the transmission of the data. Data will be transported using a flash drive, designated only for research purposes.